CLINICAL TRIAL: NCT05435092
Title: Influence of Native Knee Anatomy on Alignment and Outcome After Total Knee Arthroplasty CAT - Clinical Correlation of TKA Alignment and Native Knee Alignment
Brief Title: Clinical Correlation of TKA Alignment and Native Knee Anatomy
Acronym: CAT
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-00084; mu22Mueller
Record Dates: First submitted 2022-06-15; First posted 2022-06-28 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Total Knee Arthroplasty (TKA)
Keywords: osteoarthritis; knee protheses; knee replacement; knee alignment; knee pain; 3D-reconstruction Computer Tomography
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients scheduled for primary TKA: Adult Patients diagnosed with osteoarthritis of the knee and who are scheduled for a primary total knee arthroplasty
  Interventions: Radiation: 3D-reconstruction CT

INTERVENTIONS:
Radiation: 3D-reconstruction CT — Three dimensional CT (3D CT):Method of surface rendition of anatomy by means of a special computer software to capture 3D bone models used to improve the outcomes of Total Knee Arthroplasty (TKA).

SUMMARY:
Total knee arthroplasty (TKA) is still considered the treatment of choice for painful osteoarthritis. In the last decades neutral mechanical knee alignment in the coronal plane has been considered the gold standard. However, the optimal TKA alignment is still debated. Today, component rotation measurements on three-dimensional (3D) reconstructed computed tomography (CT) images are considered the gold standard for assessing native preoperative alignment and TKA component position. In this study pre-and postoperative radiographic measurements, functional scores, and biomechanical parameters of patients with knee osteoarthritis will be assessed with the aim to investigate the relationship between deviations of TKA alignment from native preoperative alignment and clinical, functional and biomechanical alignment.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is still considered the treatment of choice for painful osteoarthritis resulting in pain and functional improvement. Despite the development of novel prosthetic design and improved outcome, about 20% of patients report persisting pain interfering with their daily activities.Total knee prostheses are aligned in the coronal, sagittal and axial planes during implantation. In the last decades, neutral mechanical knee alignment in the coronal plane has been considered the gold standard. The aim of mechanical alignment in TKA is to achieve a femorotibial joint line that is perpendicular to the mechanical axis of the long leg axis hence correcting any varus-valgus deformity via prosthesis placement with the goal of equally distributing the load between the medial and lateral prosthesis component. However, the optimal TKA alignment is still debated. Traditionally, knee alignment and total knee arthroplasty component position have been assessed using radiographs. However, this method has a low accuracy and reliability because of variation in limb rotation, knee extension deficit, patient positioning, or magnification factors. Component rotation measurements on three-dimensional (3D) reconstructed computed tomography (CT) images have replaced former methods and are now considered the gold standard for assessing native preoperative alignment and TKA component position. In this study pre-and postoperative radiographic measurements, functional scores, and biomechanical parameters of patients with knee osteoarthritis will be assessed with the aim to investigate the relationship between deviations of TKA alignment from native preoperative alignment and clinical, functional and biomechanical alignment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosed osteoarthritis of the knee
* Planned primary total knee arthroplasty (cruciate retaining (CR) or posterior stabilizing (PS) designs)

Exclusion Criteria:

* Inability to provide informed consent
* Inability to communicate in German, French, Italian or English
* Any previous ipsilateral bony knee procedure prior to TKA
* Planned partial knee arthroplasty, semi- or full-constrained knee prosthesis
* Patients unlikely to attend clinical follow-up (e.g., when living abroad)
* Pregnancy
* Female participants of childbearing potential, not using a medically reliable method of contraception, who do not wish to undergo a pregnancy test prior to exposure to i ionizing radiation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with knee osteoarthritis who are scheduled for a primary total knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Deviation of TKA alignment from preoperative native knee alignment in the coronal plane | 3 months
  Primary radiographic endpoints to assess alignment deviations in the coronal plane:
  1. Whole limb mechanical axis (hip-knee-ankle (HKA) angle, preoperative)
  2. Native femoral varus/valgus alignment (preoperative)
  3. Native tibial varus/valgus alignment (preoperative)
  4. Femoral component varus/valgus alignment
  5. Tibial component varus/valgus alignment

SECONDARY OUTCOMES:
Evaluation of the Sagittal alignment | 3 months
  Evaluation of the
  * Flexion/extension alignment of the femur (preoperative)
  * Native tibial posterior slope (preoperative)
  * Flexion/extension alignment of the femoral component
  * Tibial component posterior slope
Evaluation of the Axial alignment | 3 months
  Evaluation of the
  * Native femoral rotation (preoperative)
  * Native tibial rotation (preoperative)
  * Rotation of the femoral component
  * Rotation of the tibial component
  * Component mismatch rotation
Assessment of Clinical, functional and biomechanical parameters | 2 years
  Functional scores:
  * Oxford Knee Score (OKS)
  * Knee Osteoarthritis Outcome Score (KOOS)
  * KSS (Knee Society Score)
  * NPRS (numeric pain rating scale)
  * EQ-5D-5L
  Biomechanical parameters:
  * Spatiotemporal parameters: walking speed, cadence, stride length, stride duration
  * Sagittal plane kinematic parameters: difference in dynamic knee flexion range of motion stance, dynamic knee flexion range of motion gait cycle and dynamic hip flexion range of motion stance between affected and unaffected leg
  * Ambulatory joint mechanics parameters: differences in 3-dimensional joint moments and medial and lateral compartment contact forces, tibia rotation, tibia translation and muscle activation patterns
  * Muscle strength: Differences in isokinetic muscle strength in knee flexion and knee extension
  Local adverse events: persistent or worsening pain; infection; any local event

OTHER OUTCOMES:
Deviation of preoperative native knee alignment from neutral alignment in the coronal plane | 3 months
  Primary radiographic endpoints to assess alignment deviations in the coronal plane:
  1. Whole limb mechanical axis (hip-knee-ankle (HKA) angle, preoperative)
  2. Native femoral varus/valgus alignment (preoperative)
  3. Native tibial varus/valgus alignment (preoperative)
  4. Femoral component varus/valgus alignment
  5. Tibial component varus/valgus alignment

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M. Müller, Prof.Dr.med., Study Director — University Hospital of Basel
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided